CLINICAL TRIAL: NCT06239441
Title: Assessment and Prediction of the Effectiveness of Mepolizumab Anti-IL-5/IL5R Inhibitors in a Real-world Setting
Brief Title: Effectiveness of Anti-IL-5/IL5R Inhibitors
Status: Completed | Type: Observational
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Catherine Lemiere, MD, MSc, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Other Study IDs: 2021-2190
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Severe Asthma
Keywords: Severe Asthma; IL5 antagonist
MeSH Terms: conditions — Asthma | interventions — mepolizumab; benralizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: IL5/IL5R Antagonists — Treatment with IL5/IL5R antagonists for one year
  Other Names: mepolizumab, benralizumab

SUMMARY:
The goal of this observational study is to assess the response to treatment, in patients 18 years and older diagnosed with severe asthma in whom an IL5/IL5R antagonists was initiated between 2012 and 2020.

The main question[s] it aims to answer are:

* What is the response rate after one year of treatment with IL5/IL5R antagonists.
* What is the response and remission rate after one year of treatment with IL5/IL5R antagonists in subjects who fullfilled the original randomized control trials (RCTs) inclusion criteria compared with those who did not.

DETAILED DESCRIPTION:
IL5/IL5-receptor (IL5R) antagonists are effective in reducing asthma exacerbations and have a corticosteroid sparing effect in selected severe eosinophilic asthmatics. The original randomized clinical trials that assessed the efficacy of IL5/IL5-R antagonists included highly selected patients who are not necessarily representative of the asthmatic population treated with IL5/IL5R antagonists in clinical practice.

The aims of this study are:

1. To assess the response to treatment, in patients 18 years and older diagnosed with severe asthma in whom an IL5/IL5R antagonists was initiated between 2012 and 2020.
2. To compare the response and remission rate after one year of treatment with IL5/IL5-R antagonists in asthmatics who would and would have not met the inclusion criteria of the original randomized clinical trials.

We will perform a retrospective cohort study using data from the hospital charts of severe asthmatics treated with mepolizumab, reslizumab or benralizumab between November 2012 and December 2020 at the outpatient asthma clinic of a tertiary center (Sacre-Coeur Hospital) in Montreal. Cohort entry (CE) will be defined as the first prescription filled of IL5/IL5R antagonists. Authorization from the research ethics committee of the CIUSSS du Nord-de-l'île-de-Montréal and from the director of Professional Services was obtained.

Statistical analysis Descriptive statistics will be used to summarize clinical, functional, and demographic characteristics of the patients of the whole cohort, as well as of the RCT in group and RCT out group. Baseline data will be recorded on the date closest to cohort entry. Results will be expressed as mean and standard deviation, except for data with a non-normal distribution, which were expressed as median and interquartile ranges and proportions for categorical variables. Chi-squared test and Student's t test will be used to compare patients' characteristics between RCT in group and RCT out group. All tests will be two-tailed, and the statistical significance level will be set at 0.05.

Logistic regression analyses will be performed to identify factors associated with a positive response to treatment as well as the achievement of remission on treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients 18 years and older diagnosed with severe asthma in whom an IL5/IL5R antagonist was initiated at the outpatient asthma clinic of a tertiary center (Sacre-Coeur Hospital) in Montreal.c between 2012 and 2020.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years and older diagnosed with severe asthma in whom an IL5/IL5R antagonist was initiated between 2012 and 2020 for were included. Data recorded in the year preceding the initiation of IL5/IL5R antagonist were compared with data recorded in the year following the initiation of the biological therapy.
  Subjects who were aged 75 years or younger, had a smoking history of less than 10 pack-year, a FEV1 of less than 80% of the predicted value along with FEV1 reversibility of at least 12% and 200 ml in the previous year were considered as fulfilling the inclusion criteria of the original RCTs (RCT in group). Subjects who did not meet one of those criteria were considered as not fulfilling the original RCT inclusion criteria (RCT out group).
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lemiere, MD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RCT in Group: Subjects who were aged 75 years or younger, had a smoking history of less than 10 pack-year, a FEV1 of less than 80% of the predicted value along with FEV1 reversibility of at least 12% and 200 ml.
- RCT Out Group: Subjects who did not meet one of those criteria:
  age 75 or younger FEV1 less than 80% FEV1 reversibility after bronchodilator of at least 12% and 200ml.
Period: Overall Study
Arm/Group | RCT in Group | RCT Out Group
Started | 22 | 86
Completed | 22 | 86
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Randomized Clinical Trial (RCT) in Group: Subjects who were aged 75 years or younger, had a smoking history of less than 10 pack-year, a forced expiratory volume in one second (FEV1) of less than 80% of the predicted value along with FEV1 reversibility of at least 12% and 200 ml.
- Randomized Clinical Trial (RCT) Out Group: Subjects who did not meet one of those criteria:
  age 75 or younger FEV1 less than 80% FEV1 reversibility after bronchodilator of at least 12% and 200ml.
- Total: Total of all reporting groups
Arm/Group | Randomized Clinical Trial (RCT) in Group | Randomized Clinical Trial (RCT) Out Group | Total
Number analyzed (Participants) | 22 | 86 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.5) | 59.6 (13.6) | 58.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 51 | 64
  Male | 9 | 35 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 22 | 86 | 108
Forced expiratory volume in one second (FEV1) pre bronchodilator (BD) [Mean (Standard Deviation); unit: Litres] | 1.63 (0.54) | 1.81 (0.86) | 1.73 (0.76)
Asthma duration [Mean (Standard Deviation); unit: years] | 25.6 (16.6) | 22.9 (18.9) | 23.8 (18.5)
Atopy [Number; unit: participants] — Atopy: positivity of at least one skin prick test to common inhalants.
  participants | 19 | 55 | 74
Daily dose of inhaled corticosteroid [Mean (Standard Deviation); unit: microgram] | 1590 (419) | 1477 (576) | 1505 (548)
Number of exacerbations in the year preceding the prescription of anti IL-5 [Mean (Standard Deviation); unit: exacerbations] | 3.1 (2.5) | 3.5 (0.9) | 3.4 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Response to IL5/IL5R Antagonist
Description: Percentage of subjects achieving response to IL5/IL5R antagonists. A response to treatment was defined as a reduction of asthma exacerbations of at least 50% or a 50% or higher reduction of the OCS doses for steroid dependant patients in the year following the initiation of an IL5/IL5R antagonist compared to the year preceding the initiation of the treatment.
Time Frame: one year
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- Randomized Clinical Trial (RCT) In Group: Subjects who would have fulfilled the inclusion criteria of the landmark clinical trials on efficacy of IL-5/IL5R antagonists.
- Randomized Clinical Trial (RCT) Out Group: Subjects who would have not fulfilled the inclusion criteria of the landmark clinical trials on efficacy of IL-5/IL5R antagonists.
Arm/Group | Randomized Clinical Trial (RCT) In Group | Randomized Clinical Trial (RCT) Out Group
Number analyzed (Participants) | 17 | 80
Percent | 76.5 [54 to 99] | 82.5 [74 to 91]

2. Primary Outcome: Remission Rate With IL5/IL5R Antagonist
Description: Percentage of subjects achieving asthma remission. Clinical remission on treatment at one year was defined as no asthma exacerbation, no treatment with oral corticosteroid and a less than 10% decrease in pre-bronchodilator FEV1 compared with baseline value.
Time Frame: one year
Measure: Number (95% Confidence Interval); unit: Percent
Groups:
- RCT In: Subjects who would have fulfilled the inclusion criteria of the landmark clinical trials on efficacy of IL-5/IL5R antagonists.
- RCT Out: Subjects who would have not fulfilled the inclusion criteria of the landmark clinical trials on efficacy of IL-5/IL5R antagonists.
Arm/Group | RCT In | RCT Out
Number analyzed (Participants) | 20 | 78
Percent | 45 [21.1 to 68.9] | 24.4 [14.6 to 34.1]

ADVERSE EVENTS:
Time Frame: Adverse event were not collected
Description: This is a retrospective chart review, adverses events were not collected.
Arm/Group | RCT in Group | RCT Out Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT06239441/Prot_SAP_000.pdf